CLINICAL TRIAL: NCT01253083
Title: Mobility Training to Improve Motor Behavior in Toddlers With or at Risk for Cerebral Palsy - A Pilot Study
Brief Title: Mobility Training to Improve Motor Behavior in Toddlers With or at Risk for Cerebral Palsy: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110037; 11-CC-0037
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-04-14

CONDITIONS: Developmental Delay; Cerebral Palsy
Keywords: Mobility; Developmental Delay; Cerebral Palsy; Early Walking; Postural Control
MeSH Terms: conditions — Learning Disabilities; Cerebral Palsy

INTERVENTIONS:
Behavioral: mobility training with dynamic body weight support

SUMMARY:
Background:

- People who have cerebral palsy often have difficulty walking and moving their legs. Cerebral palsy is sometimes not identified until a child is almost 2 years of age, which means that early motor skill development can be affected and can have repercussions for later development. Studies in adults with neurological injuries (e.g., stroke, spinal cord injury) have shown that it is important to start intensive therapy soon after the injury, and it may be true that starting intensive therapy at a young age will be helpful for children with cerebral palsy. Researchers are interested in testing the effectiveness of a special body weight support system for mobility training in young children who have or are at risk for cerebral palsy.

Objectives:

- To study the effectiveness of a mobility training program on the motor skills of young children who have or are at risk for cerebral palsy.

Eligibility:

- Children between 12 and 36 months of age who have delayed motor skills and either have been diagnosed with cerebral palsy or show evidence of spasticity or brain damage.

Design:

* This study involves two 6-week study phases: a baseline phase and a mobility training program.
* Participants will be screened with a physical examination and medical history.
* During the baseline phase, participants will have mobility testing sessions once every 2 weeks. These tests will measure motor development and ability, including ease and speed of walking.
* Participants' parents/guardians will receive a mobility sensor for the child to wear at home for at least 6 hours (awake time) to measure activity and mobility levels outside of the testing sessions.
* After 6 weeks of baseline testing, participants will have 6 weeks of mobility training for 30 minutes 3 days per week. Training will involve motor tasks with weight support, conducted by a pediatric physical therapist. Activities may include walking, climbing inclines or steps, or squatting to reach toys. All sessions will be videotaped.
* To evaluate the effects of the therapy program, participants will have testing sessions every 2 weeks.
* Parents/guardians will also complete questionnaires to provide feedback on the effectiveness of the therapy program.

DETAILED DESCRIPTION:
The purpose of this pilot study is to test the feasibility and effects of a functional mobility training program on the motor ability and physical activity of young children who are developmentally delayed and at risk for cerebral palsy (CP). The study includes a sample of 10 participants between 12-36 months of age who have at least a 4 month motor delay and are at risk for CP in a single-subject research design with repeated measures during baseline and intervention phases. Participants will have biweekly assessments during the 6 week baseline phase and the subsequent 6 week mobility training phase, followed by a final assessment after 6 weeks of treatment withdraw. Assessments and training will occur in the Functional and Applied Biomechanics (FAB) section. The mobility training program consists of three days per week of 30 minute treatment sessions using dynamic body weight support during a variety of functional motor tasks. Children will be assisted, but not limited, by the dynamic weight support system while they are encouraged to participate in a variety of age-appropriate mobility tasks. It is hypothesized that this system combined with the functional activity practice will facilitate the development of postural control and strength, and thereby improve walking ability. The primary outcome measures are completion rate and gross motor ability as measured by the Gross Motor Function Measure (GMFM). Secondary outcome measures include the amount of gross motor delay as measured by the Bayley Motor Scale (BMS),, the Functional Mobility Scale (FMS), spatiotemporal gait measures, and amount of physical activity in daily life. Results of this pilot study will be used to refine the mobility training program, evaluate the appropriateness of the selected outcome measures, and to provide preliminary data for a larger scale clinical trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 12-36 months of age
  2. greater than or equal to 4 months of gross motor delay corrected for gestational age (measured by Bayley Motor Scale)
  3. Diagnosis of bilateral spastic cerebral palsy OR neurological evidence of spasticity or brain damage
  4. Ability to pull to stand at a surface without assistance
  5. Cognitive ability to follow one-step commands
  6. Availability to return to NIH CC with parent or caregiver for required treatment and assessment sessions

EXCLUSION CRITERIA:

1. Unilateral cerebral palsy
2. Secondary orthopedic, neuromuscular or cardiovascular condition unrelated to CP
3. Greater than six months of independent walking experience
4. History of surgery or injury to the lower extremities in the past 6 months

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2010-11-15; Primary Completion 2014-06-06 (Actual); Study Completion 2014-06-06 (Actual)

PRIMARY OUTCOMES:
Change in motor delay

SECONDARY OUTCOMES:
Completion rate, change in gross motor function, change in functional mobility, change in walking speed, change in physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Yeargin-Allsopp M, Van Naarden Braun K, Doernberg NS, Benedict RE, Kirby RS, Durkin MS. Prevalence of cerebral palsy in 8-year-old children in three areas of the United States in 2002: a multisite collaboration. Pediatrics. 2008 Mar;121(3):547-54. doi: 10.1542/peds.2007-1270. PMID 18310204
- [Background] Odding E, Roebroeck ME, Stam HJ. The epidemiology of cerebral palsy: incidence, impairments and risk factors. Disabil Rehabil. 2006 Feb 28;28(4):183-91. doi: 10.1080/09638280500158422. PMID 16467053